CLINICAL TRIAL: NCT06303518
Title: Effects of End Tidal Carbon Dioxide Concentration on Depth of Anesthesia in Children Undergoing Total Intravenous Anesthesia
Brief Title: End Tidal Carbon Dioxide Concentration and Depth of Anesthesia in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Chin, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H23-03546
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Hypercapnia; Hypocapnia
MeSH Terms: conditions — Hypercapnia; Hypocapnia

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a randomized, prospective, crossover trial. The six arms will be as below:
  1. Normal ETCO2 -> High Normal ETCO2 -> Low Normal ETCO2
  2. Normal ETCO2 -> Low Normal ETCO2 -> High Normal ETCO2
  3. High Normal ETCO2 -> Low Normal ETCO2 -> Normal ETCO2
  4. High Normal ETCO2 -> Normal ETCO2 -> Low Normal ETCO2
  5. Low Normal ETCO2 -> High Normal ETCO2 -> Normal ETCO2
  6. Low Normal ETCO2 -> Normal ETCO2 -> High Normal ETCO2
Who Masked: Care Provider
Masking Description: The anesthesiologist will be blinded to the BIS reading and will continue to provide anesthesia according to the protocol. The BIS numerical value in the OR will be covered, but the waveform will be visible to assess signal quality. The anesthesiologist providing care to the patient will not be involved in data collection or analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- High normal ETCO2, Normal ETCO2, Low normal ETCO2 (Experimental): All patients will receive same interventions, in a randomised order.
  Interventions: Other: High normal ETCO2: ETCO2 50 mmHg (+/- 3mmHg); Other: Normal ETCO2: ETCO2 40 mmHg (+/- 3mmHg); Other: Low Normal ETCO2: ETCO2 30 mmHg (+/- 3mmHg)
- High normal ETCO2, Low normal ETCO2, Normal ETCO2 (Experimental): All patients will receive same interventions, in a randomised order.
  Interventions: Other: High normal ETCO2: ETCO2 50 mmHg (+/- 3mmHg); Other: Normal ETCO2: ETCO2 40 mmHg (+/- 3mmHg); Other: Low Normal ETCO2: ETCO2 30 mmHg (+/- 3mmHg)
- Low normal ETCO2, Normal ETCO2, High normal ETCO2 (Experimental): All patients will receive same interventions, in a randomised order.
  Interventions: Other: High normal ETCO2: ETCO2 50 mmHg (+/- 3mmHg); Other: Normal ETCO2: ETCO2 40 mmHg (+/- 3mmHg); Other: Low Normal ETCO2: ETCO2 30 mmHg (+/- 3mmHg)
- Low normal ETCO2, High normal ETCO2, Normal ETCO2 (Experimental): All patients will receive same interventions, in a randomised order.
  Interventions: Other: High normal ETCO2: ETCO2 50 mmHg (+/- 3mmHg); Other: Normal ETCO2: ETCO2 40 mmHg (+/- 3mmHg); Other: Low Normal ETCO2: ETCO2 30 mmHg (+/- 3mmHg)
- Normal ETCO2, Low normal ETCO2, High normal ETCO2 (Experimental): All patients will receive same interventions, in a randomised order.
  Interventions: Other: High normal ETCO2: ETCO2 50 mmHg (+/- 3mmHg); Other: Normal ETCO2: ETCO2 40 mmHg (+/- 3mmHg); Other: Low Normal ETCO2: ETCO2 30 mmHg (+/- 3mmHg)
- Normal ETCO2, High normal ETCO2, Low normal ETCO2 (Experimental): All patients will receive same interventions, in a randomised order.
  Interventions: Other: High normal ETCO2: ETCO2 50 mmHg (+/- 3mmHg); Other: Normal ETCO2: ETCO2 40 mmHg (+/- 3mmHg); Other: Low Normal ETCO2: ETCO2 30 mmHg (+/- 3mmHg)

INTERVENTIONS:
Other: High normal ETCO2: ETCO2 50 mmHg (+/- 3mmHg) — BIS readings will be recorded continuously at 'High Normal ETCO2' (50 mmHg +/- 3 mmHg). Each patient will be tested at High normal, normal, and low normal ETCO2 levels in a randomized order.
Other: Normal ETCO2: ETCO2 40 mmHg (+/- 3mmHg) — BIS readings will be recorded continuously at 'Normal ETCO2' (40 mmHg +/- 3 mmHg). Each patient will be tested at High normal, normal, and low normal ETCO2 levels in a randomized order.
Other: Low Normal ETCO2: ETCO2 30 mmHg (+/- 3mmHg) — BIS readings will be recorded continuously at 'Low Normal ETCO2' (30 mmHg +/- 3 mmHg). Each patient will be tested at High normal, normal, and low normal ETCO2 levels in a randomized order.

SUMMARY:
Carbon Dioxide (CO2) is a by-product of metabolism and is removed from the body when we breathe out. High levels of CO2 can affect the nervous system and cause us to be sleepy or sedated. Research suggests that high levels of CO2 may benefit patients who are asleep under anesthesia, such as by reducing infection rates, nausea, or recovery from anesthesia . CO2 may also reduce pain signals or the medication required to keep patients asleep during anesthesia; this has not been researched in children.

During general anesthesia, anesthesiologists keep patients asleep with anesthetic gases or by giving medications into a vein. These drugs can depress breathing; therefore, an anesthesiologist will control breathing (ventilation) with an artificial airway such as an endotracheal tube. Changes in ventilation can alter the amount of CO2 removed from the body. The anesthesiologist may also monitor a patient's level of consciousness using a 'Depth of Anesthesia Monitor' such as the Bispectral Index (BIS), which analyzes a patient's brain activity and generates a number to tell the anesthesiologist how asleep they are.

The investigator's study will test if different levels of CO2 during intravenous anesthesia are linked with different levels of sedation or sleepiness in children, as measured by BIS. If so, this could reduce the amount of anesthetic medication the child receives. Other benefits may be decreased medication costs, fewer side effects, and a positive environmental impact by using less disposable anesthesia equipment.

DETAILED DESCRIPTION:
Purpose: Carbon dioxide (CO2) is a major end-product of metabolism and can have marked effects on central nervous system function. It can also be easily manipulated during general anesthesia via controlled ventilation. High levels of carbon dioxide (hypercapnia) are associated with sedation and have been shown to produce selective suppression of thermal and ischaemic pain in animals and humans. This effect was attenuated by dexamethasone and naloxone, indicating that stress pathways and endogenous opioids may be implicated. Hypercapnia during anesthesia may have additional benefits, including reduced levels of wound infection due to improved tissue oxygenation reduced incidence of postoperative nausea and vomiting and reduced recovery time from volatile anesthetic.

It is a known phenomenon for high levels of CO2 to be associated with reduced levels of consciousness in humans, known as CO2 narcosis. A 1927 paper described narcosis of animals when breathing 30-40% CO2 in oxygen, with prompt recovery upon removal. The authors described a 'sharp sour taste' and associated hypertension when the same solution was administered to humans. However, few studies investigate the impact of carbon dioxide on anesthetic requirements. An animal study from 1967 demonstrated that very high levels of CO2 (>95 mmHg) offset halothane requirements in dogs. Most recently, increased carbon dioxide levels during surgery (40 - 45 mmHg) were shown to reduce the Minimal Alveolar Concentration to Blunt Adrenergic Response (skin incision; MAC-BAR) of sevoflurane in adult patients undergoing gastric carcinoma resection.

Total intravenous anesthesia (TIVA), an alternative to inhalational anesthesia, is a commonly used anesthetic technique in the investigator's institution. This is due to its many benefits, including reduced emergence delirium, reduced environmental impact and reduced post-operative nausea and vomiting. Administration can be guided by depth of anesthesia monitoring such as the Bispectral Index (BIS), which measures the patient's level of consciousness derived from electroencephalogram readings. BIS has been shown to help guide propofol dosing in children regardless of whether the TIVA technique was target controlled or a manual infusion regimen, and to correlate well with both modelled and measured propofol levels in children.

The investigator's study aims to determine whether differing levels of CO2 affect the anesthetic depth in anesthetized children, as measured by BIS.

Hypothesis: Hypercarbia is associated with a reduction in BIS readings, in anesthetized children.

Justification: The impact of EtCO2 on BIS has not been studied in children. If discovered, a correlation between the two could significantly change anesthetic practice. It is straightforward to increase EtCO2 levels in anesthetized patients, and if this was found to reduce their anesthetic requirements it could enable lower rates of anesthetic drug administration. This would benefit the patient by exposing them to less medication and fewer associated side effects, as well as benefitting the hospital and wider environment by reducing cost and use of disposable equipment such as ampoules, packaging and syringes.

Objectives: (1) To determine the effect of EtCO2 on the depth of anesthesia in children, as measured by BIS.

(2) Patient movement as detected clinically by the surgical or anesthetic team.

Research Design: The investigators plan to conduct a randomized, prospective, crossover trial. The within-subject design allows patients to act as their own controls. The order in which the EtCO2 levels are tested will be randomized between patients using sealed envelopes. The anesthesiologist in the room will be blinded to the BIS reading but will be informed by a research assistant if it reads persistently high (>60) for over one minute.

Statistical analysis: Physiological data will be collected in real-time using purpose-built software. Patient demographics and characteristics will be collected by a research assistant. Time-series plots of BIS and EtCO2 for each participant will be made in R (R Foundation for Statistical Computing, Vienna, Austria). Generalized estimating equations (GEE), using the geepack package, will be applied to estimate the effect of changes in target EtCO2 on serial BIS measurements during the anesthesia maintenance phase. Each participant will be considered their own data cluster to provide an appropriate grouping structure for the analysis. An independent correlation structure will be applied, and a robust (sandwich) estimator method will be used to obtain standard errors.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 - 11 years undergoing non- or minimally-stimulating elective procedures, defined as anesthesia without skin incision or painful manipulation (e.g., non-invasive imaging, auditory brainstem response testing), middle ear surgery, surgery with effective local or regional anesthesia before surgical incision (e.g dental procedures with local anesthetic infiltration, urology with regional block).
* American Society of Anesthesiologists (ASA) physical status I and II
* TIVA technique appropriate throughout induction and maintenance of anesthesia
* Controlled ventilation via endotracheal tube
* Anticipated surgical time ≥ 90 minutes: to allow time for anesthetic induction and subsequent testing and washout periods at all three EtCO2 levels.

Exclusion Criteria:

* Need for inhalational induction of anesthesia
* Sedative premedication
* Use of ketamine intraoperatively
* Unable to place BIS electrodes due to surgical site or other contraindications (e.g., MRI)
* Allergy to study drugs (propofol, remifentanil, lidocaine)
* Depression of conscious level for any reason
* BMI <5th or >95th centile for age
* History of obstructive or central sleep apnea
* Known or suspected raised intracranial pressure
* Recent or historical traumatic brain injury

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of end-tidal carbon dioxide concentration (EtCO2) on the depth of anesthesia in children, as measured by BIS. | Continually assessed throughout the general anesthetic, approximately 1.5-2 hours
  The investigator's study aims to determine whether differing levels of CO2 affect the anesthetic depth in anesthetized children, as measured by BIS. The investigators will determine a significant change in BIS to be at least a 5 point difference. Patients will act 'as their own controls', and be tested across three ETCO2 levels in a randomized order.

SECONDARY OUTCOMES:
Patient movement as detected clinically by the surgical or anesthetic team. | Continually assessed throughout the general anesthetic, approximately 1.5-2 hours
  Clinical indicators of inadequate aesthetic depth, to be recorded on data collection team if observed by any member of the clinical team.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Chin, MBBS, FRCA, FRCP, MA, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WOODBURY DM, KARLER R. The role of carbon dioxide in the nervous system. Anesthesiology. 1960 Nov-Dec;21:686-703. doi: 10.1097/00000542-196011000-00012. No abstract available. PMID 13786527
- [Background] Fukuda T, Hisano S, Toyooka H. Moderate hypercapnia-induced anesthetic effects and endogenous opioids. Neurosci Lett. 2006 Jul 31;403(1-2):20-3. doi: 10.1016/j.neulet.2006.04.026. Epub 2006 May 15. PMID 16701947
- [Background] Gronroos M, Pertovaara A. A selective suppression of human pain sensitivity by carbon dioxide: central mechanisms implicated. Eur J Appl Physiol Occup Physiol. 1994;68(1):74-9. doi: 10.1007/BF00599245. PMID 8162926
- [Background] Akca O, Liem E, Suleman MI, Doufas AG, Galandiuk S, Sessler DI. Effect of intra-operative end-tidal carbon dioxide partial pressure on tissue oxygenation. Anaesthesia. 2003 Jun;58(6):536-42. doi: 10.1046/j.1365-2044.2003.03193.x. PMID 12846617
- [Background] Saghaei M, Matin G, Golparvar M. Effects of intra-operative end-tidal carbon dioxide levels on the rates of post-operative complications in adults undergoing general anesthesia for percutaneous nephrolithotomy: A clinical trial. Adv Biomed Res. 2014 Feb 28;3:84. doi: 10.4103/2277-9175.127997. eCollection 2014. PMID 24761392
- [Background] Katznelson R, Djaiani G, Naughton F, Wasowicz M, Ragoonanan T, Duffin J, Fedorko L, Murphy J, Fisher JA. Post-operative hypercapnia-induced hyperpnoea accelerates recovery from sevoflurane anaesthesia: a prospective randomised controlled trial. Acta Anaesthesiol Scand. 2013 May;57(5):623-30. doi: 10.1111/aas.12093. Epub 2013 Mar 3. PMID 23452265
- [Background] Yamaguchi J, Kinoshita K, Hosokawa T, Ihara S. "The eyes are the windows of the soul": Portable automated pupillometry to monitor autonomic nervous activity in CO2 narcosis: A case report. Medicine (Baltimore). 2023 May 12;102(19):e33768. doi: 10.1097/MD.0000000000033768. PMID 37171322
- [Background] Leake CD, Waters RM. Leake CD, Waters RM (1928) The anaesthetic properties of carbon dioxide. J Pharmacol Exp Ther 33:280-281. In.
- [Background] Eisele JH, Eger EI 2nd, Muallem M. Narcotic properties of carbon dioxide in the dog. Anesthesiology. 1967 Sep-Oct;28(5):856-65. doi: 10.1097/00000542-196709000-00019. No abstract available. PMID 6035017
- [Background] Wu Z, Yu J, Zhang T, Tan H, Li H, Xie L, Lin W, Shen D, Cao L. Effects of Etco2 on the Minimum Alveolar Concentration of Sevoflurane that Blunts the Adrenergic Response to Surgical Incision: A Prospective, Randomized, Double-Blinded Trial. Anesth Analg. 2022 Jul 1;135(1):62-70. doi: 10.1213/ANE.0000000000005784. Epub 2022 Jun 16. PMID 34744156
- [Background] Chandler JR, Myers D, Mehta D, Whyte E, Groberman MK, Montgomery CJ, Ansermino JM. Emergence delirium in children: a randomized trial to compare total intravenous anesthesia with propofol and remifentanil to inhalational sevoflurane anesthesia. Paediatr Anaesth. 2013 Apr;23(4):309-15. doi: 10.1111/pan.12090. PMID 23464658
- [Background] Narayanan H, Raistrick C, Tom Pierce JM, Shelton C. Carbon footprint of inhalational and total intravenous anaesthesia for paediatric anaesthesia: a modelling study. Br J Anaesth. 2022 Aug;129(2):231-243. doi: 10.1016/j.bja.2022.04.022. Epub 2022 Jun 18. PMID 35729012
- [Background] Biallas R, Rusch D, de Decker W, Wulf H, Siebrecht D, Scholz J. [Prophylaxis of postoperative nausea and vomiting (PONV) in children undergoing strabismus surgery. Sevoflurane/N2O plus dimenhydrinate vs.propofol/remifentanil plus dimenhydrinate]. Anaesthesist. 2003 Jul;52(7):586-95. doi: 10.1007/s00101-003-0516-9. Epub 2003 Jun 18. German. PMID 12898043
- [Background] Marchant N, Sanders R, Sleigh J, Vanhaudenhuyse A, Bruno MA, Brichant JF, Laureys S, Bonhomme V. How electroencephalography serves the anesthesiologist. Clin EEG Neurosci. 2014 Jan;45(1):22-32. doi: 10.1177/1550059413509801. Epub 2014 Jan 10. PMID 24415399
- [Background] Louvet N, Rigouzzo A, Sabourdin N, Constant I. Bispectral index under propofol anesthesia in children: a comparative randomized study between TIVA and TCI. Paediatr Anaesth. 2016 Sep;26(9):899-908. doi: 10.1111/pan.12957. PMID 27461767
- [Background] Rigouzzo A, Khoy-Ear L, Laude D, Louvet N, Moutard ML, Sabourdin N, Constant I. EEG profiles during general anesthesia in children: A comparative study between sevoflurane and propofol. Paediatr Anaesth. 2019 Mar;29(3):250-257. doi: 10.1111/pan.13579. Epub 2019 Feb 12. PMID 30614153
- [Background] Rigouzzo A, Girault L, Louvet N, Servin F, De-Smet T, Piat V, Seeman R, Murat I, Constant I. The relationship between bispectral index and propofol during target-controlled infusion anesthesia: a comparative study between children and young adults. Anesth Analg. 2008 Apr;106(4):1109-16, table of contents. doi: 10.1213/ane.0b013e318164f388. PMID 18349180
- [Background] Jeleazcov C, Ihmsen H, Schmidt J, Ammon C, Schwilden H, Schuttler J, Fechner J. Pharmacodynamic modelling of the bispectral index response to propofol-based anaesthesia during general surgery in children. Br J Anaesth. 2008 Apr;100(4):509-16. doi: 10.1093/bja/aem408. Epub 2008 Feb 12. PMID 18270231
- [Background] McFarlan CS, Anderson BJ, Short TG. The use of propofol infusions in paediatric anaesthesia: a practical guide. Paediatr Anaesth. 1999;9(3):209-16. PMID 10320599
- [Background] Habre W, Disma N, Virag K, Becke K, Hansen TG, Johr M, Leva B, Morton NS, Vermeulen PM, Zielinska M, Boda K, Veyckemans F; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Incidence of severe critical events in paediatric anaesthesia (APRICOT): a prospective multicentre observational study in 261 hospitals in Europe. Lancet Respir Med. 2017 May;5(5):412-425. doi: 10.1016/S2213-2600(17)30116-9. Epub 2017 Mar 28. PMID 28363725
- [Background] Whitesell R, Asiddao C, Gollman D, Jablonski J. Relationship between arterial and peak expired carbon dioxide pressure during anesthesia and factors influencing the difference. Anesth Analg. 1981 Jul;60(7):508-12. PMID 6787952
- [Background] Wang F, Zhang J, Yu J, Tian M, Cui X, Wu A. Variation of bispectral index in children aged 1-12 years under propofol anesthesia: an observational study. BMC Anesthesiol. 2019 Aug 7;19(1):145. doi: 10.1186/s12871-019-0815-6. PMID 31390975
- [Background] Davidson A, Skowno J. Neuromonitoring in paediatric anaesthesia. Curr Opin Anaesthesiol. 2019 Jun;32(3):370-376. doi: 10.1097/ACO.0000000000000732. PMID 30893116